CLINICAL TRIAL: NCT05346705
Title: Effects of Newly-created Individualized Upper Airway Muscle Functional Training on Patients With OSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Wenyang Li, Associate Professor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AF-SOP-07-1.1-01
Record Dates: First submitted 2022-04-08; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Obstructive Sleep Apnea; Muscle Disorder
MeSH Terms: conditions — Sleep Apnea, Obstructive; Muscular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tongue/soft palate muscle control function training group (Experimental): In the sleep center, patients undergo a week of upper airway muscle training for 2 hours a day under the guidance of a doctor
  Interventions: Behavioral: New individualized upper airway muscle functional training
- Soft palate muscle group vocal resistance training group (Experimental): In the sleep center, patients undergo a week of upper airway muscle training for 2 hours a day under the guidance of a doctor
  Interventions: Behavioral: New individualized upper airway muscle functional training
- Simple tongue extension, cheek drumming/voice training group (Placebo Comparator): In the sleep center, patients undergo a week of upper airway muscle training for 2 hours a day under the guidance of a doctor
  Interventions: Behavioral: New individualized upper airway muscle functional training

INTERVENTIONS:
Behavioral: New individualized upper airway muscle functional training — The two groups of experimental groups were respectively performed tongue/soft palate muscle group control function training and soft palate muscle group vocal resistance training for 7 days.

SUMMARY:
Objectives: To observe the effect of newly-created individualized upper airway muscle functional training on the condition and intraday symptoms of OSA patients; to study the effect of this training method on the excitability of the genioglossus muscle cortex; to analyze the factors affecting the efficacy of upper airway training in the treatment of OSA and screening suitable population for upper airway training: Design: A randomized double-blind controlled trial. SAS 9.3 statistical software (SAS Institute, Cary, North Carolina, USA) was used to generate a random number table, and the selected patients were randomly divided into experimental group 1, experimental group 2, and control group according to the ratio of 1:1:1 with 100 cases each.

Unit: Shenyang, China Participants: Consecutive specific OSA patients, who are potential candidates for the treatment of upper airway training (n=300), will be recruited from a sleep center or respirologists, psychiatrists, otolaryngologists and dentists practicing with broad inclusion criteria (age: 20-75 years, AHI:15-50/h; BMI<40 kg/m2).

Interventions: The three groups of subjects completed 7-day functional training and control training of upper airway muscles in different modes, respectively completed polysomnography, neck circumference, Berlin questionnaire and Epworth sleepiness scale before and after training, The genioglossus myoelectric activity was measured after transcranial magnetic stimulation and the excitability of the genioglossus cortex motor center was used to determine the efficacy of different training. After regression analysis, the factors affecting the efficacy of upper airway muscle group training were analyzed to screen the OSA patient population suitable for upper airway muscle group training.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosis of OSA (AHI>15 events/h) announced by a sleep recording
* Mean oxygen saturation >90%
* Must be able to complete the training

Exclusion Criteria:

* Inability to tolerate overnight polysomnography in sleep lab
* >50% of observed sleep apneas being central
* Other sleep disorders such as insomnia, narcolepsy, chronic sleep deficiency, periodic limb movement disorder or restless legs syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Parameters Changes : Apnea Hypopnea Index (AHI) | Baseline and 1 Week
  Overnight polysomnography with Alice5 (Philips); AHI measured according to American Association of Sleep Medicine (AASM) criteria
Sleep Parameters Changes : Oxygen desaturation index (ODI) | Baseline and 1 Week
  Overnight polysomnography with Alice5 (Philips); ODI measured according to American Association of Sleep Medicine (AASM) criteria
Sleep Parameters Changes : Snoring index | Baseline and 1 Week
  Overnight polysomnography with Alice5 (Philips); Snoring index measured according to American Association of Sleep Medicine (AASM) criteria

SECONDARY OUTCOMES:
Upper Airway Muscle Strength (genioglossus) | Baseline and 1 Week
  Measurement of Genioglossus Strength Using the New Individualized Upper Airway Muscle Training Machine: Measuring Tongue Extension Strength (N)
Upper Airway Muscle Strength (Soft palate muscles) | Baseline and 1 Week
  Measuring Soft Palate Muscle Strength Using the New Personalized Upper Airway Muscle Training Machine: Measuring Soft Palate Muscle Resistant Pressure (kPa)
Quality of Life (as measured by Berlin Questionnaire) | Baseline and 1 Week
  The Berlin scale was used to assess the degree of risk of obstructive sleep apnea-hypopnea syndrome. The questionnaire consisted of 10 questions divided into 3 categories: snoring and apnea (5 questions); excessive daytime sleepiness or fatigue (3 questions); BMI>30 and history of hypertension. 2 or more positive results indicate a high risk of obstructive sleep apnea-hypopnea syndrome, which should be checked by the subjects, and then scored by the medical staff.
Cortical motor center excitability of upper airway muscle | Baseline and 1 Week
  Measured byTranscranial Magnetic Stimulation Machine (Nihon Nkohdencorp) : amplitude (mV)
Daytime sleepiness (as measured by Epworth Sleepiness Scale) | Baseline and 1 Week
  Scores on Epworth Sleepiness Scale range from range from 0 to 24, with higher scores indicating higher average sleep propensity in daily life (daytime sleepiness).

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No
Data can be requested from researchers after the experiment is over and after the paper is published